CLINICAL TRIAL: NCT03908827
Title: The Effectiveness of Bone Marrow Aspirate Concentrate (BMAC) in Patients With Severe Hip or Knee Osteoarthritis Awaiting Arthroplasty - A Randomized Controlled Trial
Brief Title: BMAC in Severe Hip or Knee Osteoarthritis Awaiting Arthroplasty
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Change of study design
Sponsor: CAPRI Clinic (Network)
Collaborators: Alberta Bone and Joint Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREBA.CTC-18-0114
Record Dates: First submitted 2019-04-07; First posted 2019-04-09 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Randomized Clinical Trial; Osteoarthritis; Hip; Knee; Bone Mineral Aspirate Concentrate
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will be blinded to treatment group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active BMAC treatment (Experimental): 60 mL of bone marrow will be aspirated from the iliac crest of each subject in the active treatment group. The bone marrow aspirate (BMA) will be centrifuged using a single spin protocol such that the red blood cells are minimized and the total nucleated and platelet cells are concentrated into a 12 mL volume of bone marrow aspirate concentrate (BMAC).
  Interventions: Biological: Bone Mineral Aspirate Concentrate (BMAC)
- Wait List Control (No Intervention): Participants will continue with their usual treatment, inclusive of medications or conservative treatments and will continue with activity guidelines as previously provided by clinical staff whilst awaiting joint arthroplasty

INTERVENTIONS:
Biological: Bone Mineral Aspirate Concentrate (BMAC) — A single BMAC injection will be performed into the arthritic joint
  Arms: Active BMAC treatment

SUMMARY:
The prevalence of severe and disabling osteoarthritis of the hip and/or knee in Albertans is high and increasing. Existing nonsurgical treatments often inadequately control symptoms. Analgesic medications are frequently poorly tolerated in seniors. In these circumstances, joint arthroplasty remains the most evidence based definitive treatment option. In Alberta, wait times for orthopedic assessment and joint arthroplasty are unacceptably long. Additionally, there is a subset of patients who would benefit from joint arthroplasty but are not candidates because they are too young or are poor surgical candidates because of medical comorbidities. There is a great need for a clinically effective and cost-effective nonsurgical treatment option for severe knee and hip osteoarthritis.

There is a growing body of published studies consistently documenting a good safety profile for Bone Marrow Aspirate Concentrate (BMAC) injections. The risks and adverse events are comparable to injection of commonly used therapeutic agents (i.e. corticosteroid and hyaluronic acid), including joint swelling (this risk may be increased if the joint was previously affected by gout), stiffness, soreness and, very rarely, infection. The emerging literature also documents promising improvements in pain relief and function.

If intra-articular BMAC injection results in safe, significant and predictable relief of pain and disability in Albertans with severe hip and/or knee osteoarthritis, BMAC could offer an expeditious and cost-effective alternative to joint arthroplasty thus shortening arthroplasty wait times. Additionally, patients with severe osteoarthritis who are unfit for arthroplasty could be offered this less invasive intervention.

The aim of this trial is to evaluate the safety and effectiveness of BMAC injection in patients with severe hip or knee osteoarthritis.

DETAILED DESCRIPTION:
This is a randomized controlled trial. In cooperation with Alberta Bone and Joint Health Institute (ABJHI), patients who have been deemed to be hip or knee joint arthroplasty candidates at the time of the initial assessment by the ABJHI musculoskeletal physician will be invited to participate. With the candidate's consent, they will be contacted by the study team, provided with additional information and an informed consent will be signed.

Participants will be randomized (by the project coordinator via computer generated simple randomization schedule) into either an active treatment (a single BMAC injection into the arthritic joint; n=75) or conservative care group (awaiting arthroplasty; n=75). The treatment group will receive their BMAC injection within 2 weeks of signing their consent form. 60 mL of bone marrow will be aspirated from the iliac crest of each subject in the active treatment group. The bone marrow aspirate (BMA) will be centrifuged using a single spin protocol such that the red blood cells are minimized and the total nucleated and platelet cells are concentrated into a 12 mL volume of bone marrow aspirate concentrate (BMAC). Two mL of BMA and BMAC will be retained for cellular analysis (total nucleated cells, platelet and hematocrit) injectate description purposes. Ten mL of BMAC will then be injected into the arthritic hip or knee. The bone marrow aspiration and joint injection will be done under local anesthesia, sterile technique and ultrasound or fluoroscopic guidance by a practitioner with ultrasound and fluoroscopy training/credentialing in an accredited Nonhospital Surgical Facility operating room in compliance with the College of Physicians and Surgeons of Alberta's (CPSA) Stem Cell Regenerative Therapy Standards. Each group will be allowed to take their usual analgesic medications (with the exception of the treatment group who will be asked to avoid NSAID intake for one week prior to and four weeks following their injection), receive their usual conservative treatments and each will be given the same activity instructions by ABJHI.

The active treatment group will be contacted by telephone within 3 days of their BMAC injection to monitor recovery and record and respond to any adverse events. Other outcome measures will be followed for 12 months (or until their joint arthroplasty surgery if prior to 12 months) and will be recorded by ABJHI who will be blinded to which treatment group the subjects are assigned. Outcome Measures will be measured in person at the time of enrollment into the study and at 6 months following post-treatment or non-treatment. At 3- and 12-months post, outcomes measures will be completed electronically or by phone. Only the assessor(s) will be blinded to the group assignment whereas the patient and the physician providing the treatment will be unblinded.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic advanced unilateral knee or hip osteoarthritis (Kellgren-Lawrence grade 3 or 4) that is inadequately controlled with conservative management including physical therapy, bracing and/or oral anti-inflammatory medications
* completed an intake assessment by a Hip and Knee Clinic of the Alberta Bone and Joint Health Institute with the musculoskeletal physician and have been deemed to be a candidate for a knee or hip arthroplasty

Exclusion Criteria:

* unable to provide informed consent
* have religious or other objections to the use of blood or blood products
* will not be available for the projected 1 year follow up period
* at the time of treatment have a systemic infection or a localized infection at the area of injection
* have thrombocytopenia or are on antiplatelet, anti-inflammatory or statin medications that cannot be stopped for 1 week prior to and for 1 month following the treatment.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Up to 12 months
  Participants will be asked to rate the average pain severity for the prior week of the affected joint using a Numeric Pain Rating Scale (McCaffery & Beebe, 1989). Participants will be asked to select the number that best represents their pain during the previous 24-hours on a scale of 0 to 10; with 0 indicating no pain and 10 indicating worst possible pain.

SECONDARY OUTCOMES:
Western Ontario and McMaster University Arthritis Index (WOMAC) | Up to 12 months
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Physical functioning questions cover everyday activities such as stair use, standing up from a sitting or lying position, standing, bending, walking, getting in and out of a car, shopping, putting on or taking off socks, lying in bed, getting in or out of a bath, sitting, and heavy and light household duties.
40 meter fast-paced walk test | Up to 12 months
  A fast-paced walking test that is timed over 4 x 10m (33 ft) for a total 40 m (132 ft)
30 second chair stand test | Up to 12 months
  The maximum number of chair stand repetitions possible in a 30 second period

OTHER OUTCOMES:
Healthcare utilization | Up to 12 months
  The number of physician and allied health professional visits relating to the treatment of joint pain in the prior month
Medication utilization | Up to 12 months
  Medications used to control symptoms of the arthritic joint in the prior week
Perceived need for joint arthroplasty: YES/NO | Up to 12 months
  "Given the problems you're having with your hip/knee at present, do you still want to have joint replacement surgery?"
Reported complications/Adverse events | Up to 12 months
  Descriptive list of any complications or adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Rob Burnham, MD, Principal Investigator — CAPRI Clinic
Locations (1):
- CAPRI Clinic, Lacombe, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iijima H, Isho T, Kuroki H, Takahashi M, Aoyama T. Effectiveness of mesenchymal stem cells for treating patients with knee osteoarthritis: a meta-analysis toward the establishment of effective regenerative rehabilitation. NPJ Regen Med. 2018 Sep 17;3:15. doi: 10.1038/s41536-018-0041-8. eCollection 2018. PMID 30245848
- [Background] Jevotovsky DS, Alfonso AR, Einhorn TA, Chiu ES. Osteoarthritis and stem cell therapy in humans: a systematic review. Osteoarthritis Cartilage. 2018 Jun;26(6):711-729. doi: 10.1016/j.joca.2018.02.906. Epub 2018 Mar 13. PMID 29544858
- [Background] Xing D, Wang Q, Yang Z, Hou Y, Zhang W, Chen Y, Lin J. Mesenchymal stem cells injections for knee osteoarthritis: a systematic overview. Rheumatol Int. 2018 Aug;38(8):1399-1411. doi: 10.1007/s00296-017-3906-z. Epub 2017 Dec 22. PMID 29273938
- [Background] Pas HI, Winters M, Haisma HJ, Koenis MJ, Tol JL, Moen MH. Stem cell injections in knee osteoarthritis: a systematic review of the literature. Br J Sports Med. 2017 Aug;51(15):1125-1133. doi: 10.1136/bjsports-2016-096793. Epub 2017 Mar 3. PMID 28258177
- [Background] Chakravarthy K, Chen Y, He C, Christo PJ. Stem Cell Therapy for Chronic Pain Management: Review of Uses, Advances, and Adverse Effects. Pain Physician. 2017 May;20(4):293-305. PMID 28535552
- [Background] Hegde V, Shonuga O, Ellis S, Fragomen A, Kennedy J, Kudryashov V, Lane JM. A prospective comparison of 3 approved systems for autologous bone marrow concentration demonstrated nonequivalency in progenitor cell number and concentration. J Orthop Trauma. 2014 Oct;28(10):591-8. doi: 10.1097/BOT.0000000000000113. PMID 24694554
- [Background] Shapiro SA, Kazmerchak SE, Heckman MG, Zubair AC, O'Connor MI. A Prospective, Single-Blind, Placebo-Controlled Trial of Bone Marrow Aspirate Concentrate for Knee Osteoarthritis. Am J Sports Med. 2017 Jan;45(1):82-90. doi: 10.1177/0363546516662455. Epub 2016 Sep 30. PMID 27566242
- [Background] Oliver K, Awan T, Bayes M. Single- Versus Multiple-Site Harvesting Techniques for Bone Marrow Concentrate: Evaluation of Aspirate Quality and Pain. Orthop J Sports Med. 2017 Aug 29;5(8):2325967117724398. doi: 10.1177/2325967117724398. eCollection 2017 Aug. PMID 28890905
- [Background] Sugaya H, Yoshioka T, Kato T, Taniguchi Y, Kumagai H, Hyodo K, Ohneda O, Yamazaki M, Mishima H. Comparative Analysis of Cellular and Growth Factor Composition in Bone Marrow Aspirate Concentrate and Platelet-Rich Plasma. Bone Marrow Res. 2018 Feb 25;2018:1549826. doi: 10.1155/2018/1549826. eCollection 2018. PMID 29682351
- [Background] Sampson S, Botto-van Bemden A, Aufiero D. Stem cell therapies for treatment of cartilage and bone disorders: osteoarthritis, avascular necrosis, and non-union fractures. PM R. 2015 Apr;7(4 Suppl):S26-S32. doi: 10.1016/j.pmrj.2015.01.023. PMID 25864657
- [Background] Centeno C, Sheinkop M, Dodson E, Stemper I, Williams C, Hyzy M, Ichim T, Freeman M. A specific protocol of autologous bone marrow concentrate and platelet products versus exercise therapy for symptomatic knee osteoarthritis: a randomized controlled trial with 2 year follow-up. J Transl Med. 2018 Dec 13;16(1):355. doi: 10.1186/s12967-018-1736-8. PMID 30545387
- [Background] Centeno CJ, Al-Sayegh H, Bashir J, Goodyear S, Freeman MD. A dose response analysis of a specific bone marrow concentrate treatment protocol for knee osteoarthritis. BMC Musculoskelet Disord. 2015 Sep 18;16:258. doi: 10.1186/s12891-015-0714-z. PMID 26385099
- [Background] Centeno C, Pitts J, Al-Sayegh H, Freeman M. Efficacy of autologous bone marrow concentrate for knee osteoarthritis with and without adipose graft. Biomed Res Int. 2014;2014:370621. doi: 10.1155/2014/370621. Epub 2014 Sep 7. PMID 25276781
- [Background] Pain: clinical manual for nursing practice Pain: clinical manual for nursing practice Margo McCaffery Alexander Beebe Mosby Yearbook UK pound17.25 0 7234 1992 2. Nurs Stand. 1994 Dec 7;9(11):55. doi: 10.7748/ns.9.11.55.s69. PMID 27527475
- [Background] Gill S, McBurney H. Reliability of performance-based measures in people awaiting joint replacement surgery of the hip or knee. Physiother Res Int. 2008 Sep;13(3):141-52. doi: 10.1002/pri.411. PMID 18697226
- [Background] Wright AA, Cook CE, Baxter GD, Dockerty JD, Abbott JH. A comparison of 3 methodological approaches to defining major clinically important improvement of 4 performance measures in patients with hip osteoarthritis. J Orthop Sports Phys Ther. 2011 May;41(5):319-27. doi: 10.2519/jospt.2011.3515. Epub 2011 Feb 18. PMID 21335930
- [Background] Sun Y, Sturmer T, Gunther KP, Brenner H. Reliability and validity of clinical outcome measurements of osteoarthritis of the hip and knee--a review of the literature. Clin Rheumatol. 1997 Mar;16(2):185-98. doi: 10.1007/BF02247849. PMID 9093802